CLINICAL TRIAL: NCT00027352
Title: A Large, Simple Trial Comparing Two Strategies for Management of Anti-Retroviral Therapy (The SMART Study)
Brief Title: A Comparison of Two Ways to Manage Anti-HIV Treatment (The SMART Study)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: CPCRA 065; SMART
Record Dates: First submitted 2001-12-04; First posted 2001-12-05 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2008-12

CONDITIONS: HIV Infections
Keywords: Physician's Practice Patterns; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to compare two ways of using anti-HIV drugs to help health care providers and patients decide how to best use anti-HIV treatments over many years. Many health care providers now treat patients with daily drugs to keep the viral load as low as possible. This approach helps patients with CD4 counts less than 200-250 cells/mm3 live longer without serious diseases. But it is not known if this is the best way to treat patients with higher CD4 counts. There is information suggesting that these patients may be able to wait to use anti-HIV drugs while CD4 counts are above 250 cells/mm3. Because this study will be carried out over several years, it will provide information on the long-term advantages and disadvantages of these two treatment strategies.

DETAILED DESCRIPTION:
Implementation of antiretroviral treatment (ART) guidelines, which emphasize maximal and durable suppression of viral load for the majority of individuals infected with HIV, has resulted in a substantial decline in morbidity and mortality. However, many asymptomatic patients are not at immediate risk of serious opportunistic diseases, the effectiveness of ART wanes over time due to HIV drug resistance, and there are short- and long-term toxicities of treatment. This motivates a comparison of two strategies: one which conserves treatments by deferring their use while the risk of opportunistic disease is low and one which aims for sustained virologic suppression, irrespective of disease risk.

In this large, long-term trial, patients will be randomly assigned to either the drug conservation (DC) or viral suppression (VS) group. Patients will be enrolled over a 3-year period and followed for an average of 7.5 years. The DC group will stop or defer ART until CD4 cell count declines to below 250 cells/mm3; they will then receive treatment to increase CD4 count to greater than 350 cells/mm3 followed by episodic ART based on CD4 cell count. The VS group will use ART to maintain viral load as low as possible, irrespective of CD4 cell count. Patients will be seen Months 1, 2, 4, 6, 8, 10, and 12, then every 4 months for data collection visits. All available ARTs, including immunomodulators, and resistance testing may be used by patients in both treatment groups. Selected subsamples of patients enrolled in the study will be followed with more intensive data collection for secondary outcomes relating to cost and health care utilization, quality of life, HIV transmission risk behaviors, and metabolic complications of treatment.

ELIGIBILITY:
Note: Enrollment into this trial was halted 01/11/06.

Inclusion Criteria:

* HIV infection
* CD4 cell count greater than 350 cells/mm3 within 45 days of study entry
* Willing to start, change, or stop antiretroviral therapy
* Acceptable methods of contraception
* Good health at the time of study entry
* Available for the study for at least 6 months
* Able, in the clinician's opinion, to comply with the protocol

Exclusion Criteria:

* Currently participating in the MDR-HIV, NvR study, or another study which is not consistent with one of the treatment groups in this study. CPCRA FIRST participants may be screened for SMART after August 8, 2005 and can be randomized into SMART on or after September 19, 2005.
* Pregnant or breast-feeding

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6000

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, MPH, Study Chair — Harlem AIDS Treatment Group, Harlem Hospital Center; James Neaton, PhD, Study Chair — CPCRA Statistcal and Data Management Center / CCBR
Locations (223):
- United States (105):
  - Kaiser Permanente-Fremont/Hayward Medical Centers, Fremont, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Los Angeles Gay and Lesbian Community Service Ctr, Los Angeles, California
  - Community Consortium / UCSF, San Francisco, California
  - Dr. Shawn Hassler, San Francisco, California
  - East Bay AIDS Ctr, San Francisco, California
  - Lawrence Goldyn, MD, San Francisco, California
  - Drs. Lichtenstein & Greenberg, Denver, Colorado
  - Western Infectious Disease Consultants, Denver, Colorado
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - McDowell Healthcare Center, Denver, Colorado
  - Yale U / New Haven Med Ctr / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Veterans Administration Medical Center, New Haven, Connecticut
  - Christiana Care Health Services HIV Program George, Wilmington, Delaware
  - Timothy A Price, Washington D.C., District of Columbia
  - George Washington Univ, Washington D.C., District of Columbia
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - Miami Veterans Affairs Med Ctr, Miami, Florida
  - Center for Prevention and Treatment of Infections, Pensacola, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Absolute Care Clinic, Atlanta, Georgia
  - AID Atlanta/Morehouse Med School Ryan White Cl, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta (ARCA) Central, Atlanta, Georgia
  - Cobb-Douglas County Infectious Disease Clinic, Atlanta, Georgia
  - Dekalb County Health Dept Infectious Disease, Atlanta, Georgia
  - Dr. Dennis Melton (Private Practice), Atlanta, Georgia
  - Dr. Melanie Thompson and Dr. Annette Bernard (Private Practice), Atlanta, Georgia
  - Dr. Richard Hudson (Private Practice), Atlanta, Georgia
  - HIV Services Clinic/Family Practice Medical Center, Boise, Idaho
  - Cook County Hosp, Chicago, Illinois
  - Klein and Slotten Associates / AIDS Research Alliance, Chicago, Illinois
  - Lakeshore Infectious Disease Associates, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Northside Family Medicine, Chicago, Illinois
  - Northwestern Memorial Physicians, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Southern Illinois University (SIU) School of Medicine, Springfield, Illinois
  - KU Medical School-Wichita, Midtown Clinic, Wichita, Kansas
  - KU Medical School-Wichita, MPA, Wichita, Kansas
  - University of Mississippi Medical Center, New Orleans, Louisiana
  - Our Lady of the Lake Regional Med Ctr, New Orleans, Louisiana
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Community Research Initiatives of New England, Boston, Massachusetts
  - Community Research Initiatives/ProACT, Boston, Massachusetts
  - Community Research Initiative/ProACT, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Detroit Community Health Connection, Detroit, Michigan
  - Detroit Receiving, Detroit, Michigan
  - Wayne State Univ / Medical College of Ohio at Toledo, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Mt. Clemens General Hospital, Detroit, Michigan
  - Providence Hosp- Newland Med Assoc. Inc., Detroit, Michigan
  - McAuley Health Center, Grand Rapids, Michigan
  - Michigan State University Infectious Diseases Clinic, Lansing, Michigan
  - William Beaumont Hospital/CORNET, Royal Oak, Michigan
  - Mayo Clinic/CORNET, Rochester, Minnesota
  - Cooper Hospital Early Intervention Program, Camden, New Jersey
  - Jersey Shore Med Ctr, Neptune City, New Jersey
  - Raritan Bay Med Ctr, Newark, New Jersey
  - Saint Michael's Med Ctr, Newark, New Jersey
  - Jeffrey Bomser Clinic / NJCR, Newark, New Jersey
  - New Jersey Community Research Initiative, Newark, New Jersey
  - NJCRI, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Poinnt, New Jersey
  - SUNY Downstate Med Ctr, Brooklyn, New York
  - Grant Houses Health Ctr, New York, New York
  - HHC MMC Unit #1, New York, New York
  - HHC Outpatient Clinics, New York, New York
  - Jacobi Medical Center, New York, New York
  - Lenox Avenue Health Ctr, New York, New York
  - Lincoln Medical & Mental Health Center, New York, New York
  - Polo Grounds Health Care Ctr, New York, New York
  - Syndenham Neighborhood Family Care Ctr, New York, New York
  - Metropolitan Hospital Center, New York, New York
  - Bronx-Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Veterans Affairs Medical Center, The Bronx, New York
  - Wake Forest Univ Health Sciences, Winston-Salem, North Carolina
  - Univ of Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - Legacy Clinic NE, Portland, Oregon
  - Salem Hospital, Portland, Oregon
  - The Research & Education Group / Multomah Cnty Hlth Dept, Portland, Oregon
  - The Research & Education Group / The R & E Grp Office, Portland, Oregon
  - The Research & Education Grp / Oregon Hlth Sci Univ, Portland, Oregon
  - The Rsch & Ed Grp / Legacy Cln at Good Samaritan, Portland, Oregon
  - The Rsch & Ed Grp / Providence Portland Med Ctr, Portland, Oregon
  - The Research and Education Group, Portland, Oregon
  - Penn Community Infectious Diseases, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Temple Univ School of Medicine, Philadelphia, Pennsylvania
  - Montrose Clinic, Houston, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas
  - University Clinical Research Center, Houston, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Infectious Disease Associates of Virginia, Lynchburg, Virginia
  - Cross Over Clinic / Div of Infectious Diseases, Richmond, Virginia
  - McGuire VA / Division of Infectious Diseases, Richmond, Virginia
  - MCV ID Clinic, Richmond, Virginia
  - MediCorp, Infectious Disease Associates, Richmond, Virginia
  - Petersburg Health Care Alliance, Richmond, Virginia
  - South Richmond Health Ctr, Richmond, Virginia
  - Vernon J. Harris East End Community Health Care Ct, Richmond, Virginia
  - University Of Wisconsin Hospital and Clinics/CORNET, HIV Care Program, Madison, Wisconsin
- Argentina (9):
  - Hospital de Clinicas Jose de San Martin, Buenos Aires
  - Hospital de Infecciosas F.J. Muniz, Buenos Aires
  - Hospital Gn'l de Agudos JM Ramos Mejia, Buenos Aires
  - Hospital Gn'l de Agudos T. Alvarez, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Rawson, Córdoba
  - Hospital Interzonall de San Juan de Dios, La Plata
  - Hospital Central, Mendoza
  - CAICI, Rosario
- Australia (8):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Prahran Market Clinic, South Yarra, Victoria
  - The Centre Clinic, South Yarra, Victoria
  - Burwood Street General Pratice, Burwood Nsw
  - Royal Perth Hosp, Perth
  - Alfred Hosp, Prahan
  - Royal Prince Alfred Hospital, Prahan
  - National Centre in HIV Epidemiology and Clinical Research, Sydney
- University of Vienna Medical School, AKH, Vienna, Austria
- Belgium (2):
  - Institute of Tropical Medicine, Antwerp
  - Centre Hospitalier Universitaire Sart-Tilman, Liège
- Brazil (12):
  - Hospital Escola Sao Francisco de Asis, Rio de Janeiro, Rio de Janeiro
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto de Infectologia Emilio Ribas, São Paulo, S.P. CEP
  - Cassiano Antonio de Moraes University Hospital, Boqueirao-Santos
  - Centro de Pesquisa Clinical do Hospital Guilherme, Boqueirao-Santos
  - Hospital de Clinicas de Porto Alegre, Porto Alegre-RS Cep
  - Hospital dos Servidores do Estado, Rio de Janeiro
  - Hospital Universitario Professor Edgard Santos, Salvador-BA
  - Ambulatorio de Imunodeficiencias Secundarias/Der30, São Paulo
  - Universidade Federal De Sao Paulo-Hospital Sao Paulo, São Paulo
  - Centro de Referencia e Treinamento DST/AIDS, São Paulo
  - Unidade de Pesquisa Clinica, São Paulo
- Canada (13):
  - Downtown Infectious Disease Clinic, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The HAVEN Program, HRSRH, Greater Sudbury, Ontario
  - Hamilton Health Science Centre-McMaster, Hamilton, Ontario
  - St. Joseph's Health Care Centre of London, London, Ontario
  - St. Josephs Hospital, London, Ontario
  - Tronto General Hospital, Toronto, Ontario
  - HIV Care Program, Windsor Regional Hospital, Windsor, Ontario
  - University de Sherbrooke, Fleurimont, Quebec
  - Clinique Medicale L'actuel, Montreal, Quebec
  - Montreal Chest Institute/Royal Victoria Hospital, Montreal, Quebec
  - Centre hospitalier de l'universite Laval (CHUL), Sainte-Foy, Quebec
  - Recherche Clinique Centre Medical Halles de Saint-, Ste-Foy, Quebec
- West-Tallinn Central Hospital, Tallinn, Estonia
- France (7):
  - CHU de la Region Annecienne, Annecy
  - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire, Chu-grenoble
  - Hopital Louis Mourier, Colombes
  - Hopital Sainte-Marguerite, Marseille
  - Hopital Saint-Louis, Paris
  - Hopital Pitie Salpetriere, Paris
- Germany (4):
  - Klinik fur Dermatologie, Venerologie, Allergologie, Essen
  - Johann Wolfgang Goethe University Hospital, Frankfurt am Main
  - Klinikum der Ruprecht-Karis-Universitat (U. Hospital), Heidelberg
  - University Hospital Zurich, Zurich Ch-
- St. James Hospital, Dublin, Ireland
- Ramathibodi Hospital, Tel Aviv, Israel
- Italy (10):
  - U.O. Malattie Infettive, H.S.Maria Annunziata, Antella-Firenze
  - SOCDU Malattie Infettive Ospedale Civile Asti, Asti
  - Instituto de Malattie Infettive e Tropicali, Brescia
  - Malattie Infettive Busto, Busto Arsizio (va)
  - Universita degli Studi di Modena e Reggio Emilia, Modena
  - Clinica Malattie Infettive, Pavia
  - I.R.C.C.S."L.Spallanzani", Rome
  - University of Turin, Torino
  - Servizio Regionale di Immunologia Clinica e Tipizz, Torrette Di Ancona
  - S.S. Giovanni e Paolo Hospital, Venice
- Japan (2):
  - AIDS Medical Center, International Medical Center, Tokyo
  - International Medical Center of Japan, Tokyo
- Lithuanian AIDS center, Vilnius, Lithuania
- Centre Hospitalier de Luxembourg, Barble, Luxembourg
- C.H.U. Fort-de-France, Fort-de-France, Martinique
- New Zealand (2):
  - Christchurch Hosp, Christchurch
  - Wellington Hosp, Wellington
- Ulleval Hospital, Oslo, Norway
- Peru (2):
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
- Wroclaw University School of Medicine, Koszarowa Str. 5, Poland
- Instituto A. Z. de Pesquisa e Ensino, Curitiba, Puerto Rico
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Principe de Asturias, Madrid
  - Hospital U. Virgen del Rocio, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Switzerland (5):
  - University Hospital Basel, Basel Ch
  - Poliklinik fur Infektiologie, Bern
  - Hopital de la Ville, La Chaux-de-Fonds
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Ospedale Regionale di Lugano, Lugano
- Thailand (2):
  - Sanpatong Hospital, Chiang Mai
  - Bamrasnaradura Institute, Nonthaburi
- United Kingdom (24):
  - John Radcliffe Hospital, Oxford, England
  - Royal Victoria Hospital, Belfast
  - Hawthorn House, Birmingham Heartlands NHS Trust, Birmingham
  - Southmead Hospital, Bristol
  - St. Helier Hospital, Carshalton
  - St. Helier Hospital, Carshalton, Surrey
  - Essex County Hospital, Essex
  - Victoria General Hospital, Q.E. II Health Sciences, Halifax
  - Homerton University Hospital NHS Foundation Trust, London
  - Barts and The London, NHS Trust, London
  - Central Middlesex Hospital, London
  - Royal Free Hospital, London
  - St. Thomas' Hospital, London
  - T1 Coleridge Unit, North Middlesex Hospital, London
  - The Caldecot Centre, Kings College Hospital NHS Tr, London
  - Chelsea and Westminster Hospital, London
  - St. George's Hospital, London
  - St. Mary's Hospital, London
  - The Mortimer Market Center, London
  - The James Cook University Hospital, Middlesbrough
  - Pasteur Suite, Ealing Hospital, Middlesex
  - Newcastle General Hospital, Newcastle
  - Dept. of Infection and Tropical Medicine - Royal Hallamshire Hospital, Sheffield
  - Watford Sexual Health Center;Watford General Hosp, Watford Wd

REFERENCES:
- [Background] Lederman MM, Valdez H. Immune restoration with antiretroviral therapies: implications for clinical management. JAMA. 2000 Jul 12;284(2):223-8. doi: 10.1001/jama.284.2.223. PMID 10889597
- [Background] Carpenter CC, Cooper DA, Fischl MA, Gatell JM, Gazzard BG, Hammer SM, Hirsch MS, Jacobsen DM, Katzenstein DA, Montaner JS, Richman DD, Saag MS, Schechter M, Schooley RT, Thompson MA, Vella S, Yeni PG, Volberding PA. Antiretroviral therapy in adults: updated recommendations of the International AIDS Society-USA Panel. JAMA. 2000 Jan 19;283(3):381-90. doi: 10.1001/jama.283.3.381. PMID 10647802
- [Background] Mocroft A, Katlama C, Johnson AM, Pradier C, Antunes F, Mulcahy F, Chiesi A, Phillips AN, Kirk O, Lundgren JD. AIDS across Europe, 1994-98: the EuroSIDA study. Lancet. 2000 Jul 22;356(9226):291-6. doi: 10.1016/s0140-6736(00)02504-6. PMID 11071184
- [Background] Tebas P, Henry K, Mondy K, Deeks S, Valdez H, Cohen C, Powderly WG. Effect of prolonged discontinuation of successful antiretroviral therapy on CD4+ T cell decline in human immunodeficiency virus-infected patients: implications for intermittent therapeutic strategies. J Infect Dis. 2002 Sep 15;186(6):851-4. doi: 10.1086/342603. Epub 2002 Aug 28. PMID 12198623
- [Background] Yerly S, Kaiser L, Perneger TV, Cone RW, Opravil M, Chave JP, Furrer H, Hirschel B, Perrin L. Time of initiation of antiretroviral therapy: impact on HIV-1 viraemia. The Swiss HIV Cohort Study. AIDS. 2000 Feb 18;14(3):243-9. doi: 10.1097/00002030-200002180-00006. PMID 10716500
- [Derived] Borges AH, Neuhaus J, Sharma S, Neaton JD, Henry K, Anagnostou O, Staub T, Emery S, Lundgren JD; INSIGHT SMART; START Study Groups. The Effect of Interrupted/Deferred Antiretroviral Therapy on Disease Risk: A SMART and START Combined Analysis. J Infect Dis. 2019 Jan 7;219(2):254-263. doi: 10.1093/infdis/jiy442. PMID 30032171
- [Derived] Castillo-Mancilla JR, Phillips AN, Neaton JD, Neuhaus J, Collins S, Mannheimer S, Pett S, Touzeau-Romer V, Polizzotto MN, Lundgren JD, Gardner EM; INSIGHT SMART Study Group. Association of Suboptimal Antiretroviral Therapy Adherence With Inflammation in Virologically Suppressed Individuals Enrolled in the SMART Study. Open Forum Infect Dis. 2017 Dec 22;5(1):ofx275. doi: 10.1093/ofid/ofx275. eCollection 2018 Jan. PMID 29362724
- [Derived] Larson GS, Carey C, Grarup J, Hudson F, Sachi K, Vjecha MJ, Gordin F; INSIGHT Group. Lessons learned: Infrastructure development and financial management for large, publicly funded, international trials. Clin Trials. 2016 Apr;13(2):127-36. doi: 10.1177/1740774515625974. Epub 2016 Feb 8. PMID 26908541
- [Derived] Nordell AD, McKenna M, Borges AH, Duprez D, Neuhaus J, Neaton JD; INSIGHT SMART, ESPRIT Study Groups; SILCAAT Scientific Committee. Severity of cardiovascular disease outcomes among patients with HIV is related to markers of inflammation and coagulation. J Am Heart Assoc. 2014 May 28;3(3):e000844. doi: 10.1161/JAHA.114.000844. PMID 24870935
- [Derived] Lucas GM, Cozzi-Lepri A, Wyatt CM, Post FA, Bormann AM, Crum-Cianflone NF, Ross MJ; INSIGHT SMART Study Group. Glomerular filtration rate estimated using creatinine, cystatin C or both markers and the risk of clinical events in HIV-infected individuals. HIV Med. 2014 Feb;15(2):116-23. doi: 10.1111/hiv.12087. Epub 2013 Sep 11. PMID 24024499
- [Derived] Baker JV, Brummel-Ziedins K, Neuhaus J, Duprez D, Cummins N, Dalmau D, DeHovitz J, Lehmann C, Sullivan A, Woolley I, Kuller L, Neaton JD, Tracy RP; INSIGHT SMART Study Team. HIV replication alters the composition of extrinsic pathway coagulation factors and increases thrombin generation. J Am Heart Assoc. 2013 Jul 29;2(4):e000264. doi: 10.1161/JAHA.113.000264. PMID 23896681
- [Derived] Hoy J, Grund B, Roediger M, Ensrud KE, Brar I, Colebunders R, Castro ND, Johnson M, Sharma A, Carr A; INSIGHT SMART Body Composition Substudy Group. Interruption or deferral of antiretroviral therapy reduces markers of bone turnover compared with continuous therapy: The SMART body composition substudy. J Bone Miner Res. 2013 Jun;28(6):1264-74. doi: 10.1002/jbmr.1861. PMID 23299909
- [Derived] Zetterberg E, Neuhaus J, Baker JV, Somboonwit C, Llibre JM, Palfreeman A, Chini M, Lundgren JD; INSIGHT SMART Study Group. Platelet count kinetics following interruption of antiretroviral treatment. AIDS. 2013 Jan 2;27(1):59-68. doi: 10.1097/QAD.0b013e32835a104d. PMID 23018440
- [Derived] Mocroft A, Neuhaus J, Peters L, Ryom L, Bickel M, Grint D, Koirala J, Szymczak A, Lundgren J, Ross MJ, Wyatt CM; INSIGHT SMART Study Group; ESPRIT Study Group. Hepatitis B and C co-infection are independent predictors of progressive kidney disease in HIV-positive, antiretroviral-treated adults. PLoS One. 2012;7(7):e40245. doi: 10.1371/journal.pone.0040245. Epub 2012 Jul 20. PMID 22911697
- [Derived] Baker JV, Neuhaus J, Duprez D, Cooper DA, Hoy J, Kuller L, Lampe FC, Liappis A, Friis-Moller N, Otvos J, Paton NI, Tracy R, Neaton JD; INSIGHT SMART Study Group. Inflammation predicts changes in high-density lipoprotein particles and apolipoprotein A1 following initiation of antiretroviral therapy. AIDS. 2011 Nov 13;25(17):2133-42. doi: 10.1097/QAD.0b013e32834be088. PMID 21857489
- [Derived] Mocroft A, Lifson AR, Touloumi G, Neuhaus J, Fox Z, Palfreeman A, Vjecha MJ, Hodder S, De Wit S, Lundgren JD, Phillips AN; INSIGHT SMART Study Group. Haemoglobin and anaemia in the SMART study. Antivir Ther. 2011;16(3):329-37. doi: 10.3851/IMP1746. PMID 21555815
- [Derived] Duprez DA, Neuhaus J, Tracy R, Kuller LH, Deeks SG, Orkin C, Stoehr A, Woolley IJ, Neaton JD; INSIGHT SMART Group. N-terminal-proB-type natriuretic peptide predicts cardiovascular disease events in HIV-infected patients. AIDS. 2011 Mar 13;25(5):651-7. doi: 10.1097/QAD.0b013e32834404a1. PMID 21245726
- [Derived] Lampe FC, Duprez DA, Kuller LH, Tracy R, Otvos J, Stroes E, Cooper DA, Hoy J, Paton NI, Friis-Moller N, Neuhaus J, Liappis AP, Phillips AN; INSIGHT SMART Study Group. Changes in lipids and lipoprotein particle concentrations after interruption of antiretroviral therapy. J Acquir Immune Defic Syndr. 2010 Jul;54(3):275-84. doi: 10.1097/qai.0b013e3181d32158. PMID 20658749
- [Derived] Dore GJ, Soriano V, Rockstroh J, Kupfer B, Tedaldi E, Peters L, Neuhaus J, Puoti M, Klein MB, Mocroft A, Clotet B, Lundgren JD; SMART INSIGHT study group. Frequent hepatitis B virus rebound among HIV-hepatitis B virus-coinfected patients following antiretroviral therapy interruption. AIDS. 2010 Mar 27;24(6):857-65. doi: 10.1097/QAD.0b013e328334bddb. PMID 20216301
- [Derived] Rodger AJ, Fox Z, Lundgren JD, Kuller LH, Boesecke C, Gey D, Skoutelis A, Goetz MB, Phillips AN; INSIGHT Strategies for Management of Antiretroviral Therapy (SMART) Study Group. Activation and coagulation biomarkers are independent predictors of the development of opportunistic disease in patients with HIV infection. J Infect Dis. 2009 Sep 15;200(6):973-83. doi: 10.1086/605447. PMID 19678756
- [Derived] Grund B, Peng G, Gibert CL, Hoy JF, Isaksson RL, Shlay JC, Martinez E, Reiss P, Visnegarwala F, Carr AD; INSIGHT SMART Body Composition Substudy Group. Continuous antiretroviral therapy decreases bone mineral density. AIDS. 2009 Jul 31;23(12):1519-29. doi: 10.1097/QAD.0b013e32832c1792. PMID 19531929
- [Derived] Duprez DA, Kuller LH, Tracy R, Otvos J, Cooper DA, Hoy J, Neuhaus J, Paton NI, Friis-Moller N, Lampe F, Liappis AP, Neaton JD; INSIGHT SMART Study Group. Lipoprotein particle subclasses, cardiovascular disease and HIV infection. Atherosclerosis. 2009 Dec;207(2):524-9. doi: 10.1016/j.atherosclerosis.2009.05.001. Epub 2009 May 13. PMID 19515371
- [Derived] Mocroft A, Wyatt C, Szczech L, Neuhaus J, El-Sadr W, Tracy R, Kuller L, Shlipak M, Angus B, Klinker H, Ross M; INSIGHT SMART Study Group. Interruption of antiretroviral therapy is associated with increased plasma cystatin C. AIDS. 2009 Jan 2;23(1):71-82. doi: 10.1097/QAD.0b013e32831cc129. PMID 19050388
- [Derived] Fox Z, Phillips A, Cohen C, Neuhaus J, Baxter J, Emery S, Hirschel B, Hullsiek KH, Stephan C, Lundgren J; SMART Study Group. Viral resuppression and detection of drug resistance following interruption of a suppressive non-nucleoside reverse transcriptase inhibitor-based regimen. AIDS. 2008 Nov 12;22(17):2279-89. doi: 10.1097/QAD.0b013e328311d16f. PMID 18981767
- [Derived] Tedaldi E, Peters L, Neuhaus J, Puoti M, Rockstroh J, Klein MB, Dore GJ, Mocroft A, Soriano V, Clotet B, Lundgren JD; SMART Study Group and International Network for Strategic Initiatives in Global HIV Trials (INSIGHT). Opportunistic disease and mortality in patients coinfected with hepatitis B or C virus in the strategic management of antiretroviral therapy (SMART) study. Clin Infect Dis. 2008 Dec 1;47(11):1468-75. doi: 10.1086/593102. PMID 18959492
- [Derived] Kuller LH, Tracy R, Belloso W, De Wit S, Drummond F, Lane HC, Ledergerber B, Lundgren J, Neuhaus J, Nixon D, Paton NI, Neaton JD; INSIGHT SMART Study Group. Inflammatory and coagulation biomarkers and mortality in patients with HIV infection. PLoS Med. 2008 Oct 21;5(10):e203. doi: 10.1371/journal.pmed.0050203. PMID 18942885
- [Derived] SMART Study Group; El-Sadr WM, Grund B, Neuhaus J, Babiker A, Cohen CJ, Darbyshire J, Emery S, Lundgren JD, Phillips A, Neaton JD. Risk for opportunistic disease and death after reinitiating continuous antiretroviral therapy in patients with HIV previously receiving episodic therapy: a randomized trial. Ann Intern Med. 2008 Sep 2;149(5):289-99. doi: 10.7326/0003-4819-149-5-200809020-00003. PMID 18765698
- [Derived] Strategies for Management of Anti-Retroviral Therapy/INSIGHT; DAD Study Groups. Use of nucleoside reverse transcriptase inhibitors and risk of myocardial infarction in HIV-infected patients. AIDS. 2008 Sep 12;22(14):F17-24. doi: 10.1097/QAD.0b013e32830fe35e. PMID 18753925
- [Derived] Gordin FM, Roediger MP, Girard PM, Lundgren JD, Miro JM, Palfreeman A, Rodriguez-Barradas MC, Wolff MJ, Easterbrook PJ, Clezy K, Slater LN. Pneumonia in HIV-infected persons: increased risk with cigarette smoking and treatment interruption. Am J Respir Crit Care Med. 2008 Sep 15;178(6):630-6. doi: 10.1164/rccm.200804-617OC. Epub 2008 Jul 10. PMID 18617640
- [Derived] Phillips AN, Carr A, Neuhaus J, Visnegarwala F, Prineas R, Burman WJ, Williams I, Drummond F, Duprez D, Belloso WH, Goebel FD, Grund B, Hatzakis A, Vera J, Lundgren JD. Interruption of antiretroviral therapy and risk of cardiovascular disease in persons with HIV-1 infection: exploratory analyses from the SMART trial. Antivir Ther. 2008;13(2):177-87. doi: 10.1177/135965350801300215. PMID 18505169
- [Derived] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; Lundgren JD, Babiker A, El-Sadr W, Emery S, Grund B, Neaton JD, Neuhaus J, Phillips AN. Inferior clinical outcome of the CD4+ cell count-guided antiretroviral treatment interruption strategy in the SMART study: role of CD4+ Cell counts and HIV RNA levels during follow-up. J Infect Dis. 2008 Apr 15;197(8):1145-55. doi: 10.1086/529523. PMID 18476293
- [Derived] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; Emery S, Neuhaus JA, Phillips AN, Babiker A, Cohen CJ, Gatell JM, Girard PM, Grund B, Law M, Losso MH, Palfreeman A, Wood R. Major clinical outcomes in antiretroviral therapy (ART)-naive participants and in those not receiving ART at baseline in the SMART study. J Infect Dis. 2008 Apr 15;197(8):1133-44. doi: 10.1086/586713. PMID 18476292
- [Derived] Carr A, Grund B, Neuhaus J, El-Sadr WM, Grandits G, Gibert C, Prineas RJ; SMART Study Investigators. Asymptomatic myocardial ischaemia in HIV-infected adults. AIDS. 2008 Jan 11;22(2):257-67. doi: 10.1097/QAD.0b013e3282f20a77. PMID 18097228
- [Derived] Burman WJ, Grund B, Roediger MP, Friedland G, Darbyshire J, Wu AW; SMART Study Group. The impact of episodic CD4 cell count-guided antiretroviral therapy on quality of life. J Acquir Immune Defic Syndr. 2008 Feb 1;47(2):185-93. doi: 10.1097/QAI.0b013e31815acaa4. PMID 17971716
- [Derived] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; El-Sadr WM, Lundgren J, Neaton JD, Gordin F, Abrams D, Arduino RC, Babiker A, Burman W, Clumeck N, Cohen CJ, Cohn D, Cooper D, Darbyshire J, Emery S, Fatkenheuer G, Gazzard B, Grund B, Hoy J, Klingman K, Losso M, Markowitz N, Neuhaus J, Phillips A, Rappoport C. CD4+ count-guided interruption of antiretroviral treatment. N Engl J Med. 2006 Nov 30;355(22):2283-96. doi: 10.1056/NEJMoa062360. PMID 17135583